CLINICAL TRIAL: NCT07030140
Title: A Phase II, Single-arm, Prospective Clinical Study of Neoadjuvant Therapy With Tislelizumab Combined With Radiotherapy and Gemcitabine-Platinum Chemotherapy for Borderline Resectable or Unresectable Hilar Cholangiocarcinoma
Brief Title: Phase II Study of Neoadjuvant Tislelizumab Plus Radiotherapy and GP Chemotherapy for Borderline/Unresectable Hilar Cholangiocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinbo Yue (Other)
Responsible Party: Sponsor-Investigator, Jinbo Yue, Chief Physician, Radiation Oncology, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-364-03
Record Dates: First submitted 2025-06-11; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Cholangiocarcinoma; Hilar Cholangiocarcinoma; Bile Duct Cancer
Keywords: Borderline Resectable; Unresectable; SBRT; Tislelizumab; Gemcitabine; Cisplatin; Oxaliplatin; Neoadjuvant Therapy; Immunotherapy; Radiation Therapy; PD-1 Inhibitor; Biliary Tract Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor; Bile Duct Neoplasms; Biliary Tract Neoplasms | interventions — Radiosurgery; tislelizumab; Gemcitabine; Cisplatin; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Single-arm design with sequential SBRT followed by Tislelizumab plus GP chemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab + SBRT + GP Chemotherapy (Experimental): Participants will receive neoadjuvant stereotactic body radiotherapy (SBRT) followed by three cycles of combination therapy with tislelizumab and GP chemotherapy.
  SBRT: 5 Gy × 5-8 fractions or 4 Gy × 15 fractions to the primary tumor. Tislelizumab: 200 mg intravenously every 3 weeks (Day 1 of each cycle). Gemcitabine: 1000 mg/m² IV on Days 1 and 8 of each 21-day cycle. Cisplatin: 25 mg/m² IV on Days 1 and 8 OR Oxaliplatin: 100 mg/m² IV on Day 1 (based on clinical condition). After three cycles, patients will undergo re-evaluation. Those deemed resectable will undergo surgery and receive postoperative therapy based on multidisciplinary assessment. Patients remaining unresectable will receive an additional three cycles of the same systemic therapy.
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT); Drug: Tislelizumab; Drug: Gemcitabine; Drug: Cisplatin or Oxaliplatin

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) — SBRT to the primary tumor and metastatic lymph node at a dose of either 5 Gy × 5-8 fractions or 4 Gy × 15 fractions, delivered prior to systemic therapy.
Drug: Tislelizumab — Tislelizumab 200 mg administered intravenously every 3 weeks (on Day 1 of each 21-day cycle), for three to six cycles depending on surgical eligibility.
Drug: Gemcitabine — Gemcitabine 1000 mg/m² administered intravenously on Days 1 and 8 of each 21-day cycle, for three to six cycles.
Drug: Cisplatin or Oxaliplatin — Cisplatin 25 mg/m² on Days 1 and 8 or oxaliplatin 100 mg/m² on Day 1 of each 21-day cycle, selected based on patient condition, for three to six cycles.

SUMMARY:
This is a phase II, single-arm, prospective clinical trial designed to evaluate the efficacy and safety of neoadjuvant therapy combining stereotactic body radiotherapy (SBRT), GP chemotherapy (gemcitabine and cisplatin/oxaliplatin), and tislelizumab in patients with borderline resectable or unresectable hilar cholangiocarcinoma. Eligible patients will receive SBRT followed by three cycles of tislelizumab plus GP chemotherapy. Patients with resectable disease after evaluation may undergo surgery and receive postoperative treatment as recommended by the multidisciplinary team. Those who remain unresectable will receive three additional cycles of systemic therapy. The primary endpoint is overall survival (OS); secondary endpoints include R0 resection rate, pathological complete response (pCR), surgical difficulty, progression-free survival (PFS), local control rate, and treatment-related safety.

DETAILED DESCRIPTION:
Hilar cholangiocarcinoma is a rare but highly aggressive malignancy, often diagnosed at advanced stages due to its asymptomatic progression and challenging anatomical location. R0 resection remains the cornerstone of curative therapy, but many patients are initially considered borderline resectable or unresectable due to vascular involvement or lymph node metastasis.

Recent studies suggest that neoadjuvant therapy may improve resectability and survival outcomes by reducing tumor burden and modulating the tumor microenvironment. Stereotactic body radiotherapy (SBRT) offers precise local control, while GP chemotherapy (gemcitabine and cisplatin/oxaliplatin) has demonstrated efficacy in biliary tract cancers. Immunotherapy with PD-1 inhibitors, such as tislelizumab, has shown promise in enhancing antitumor immunity, especially when combined with radiotherapy and chemotherapy.

This phase II, single-arm, prospective study aims to evaluate the efficacy and safety of neoadjuvant SBRT followed by tislelizumab and GP chemotherapy in patients with borderline resectable or unresectable hilar cholangiocarcinoma. Patients will first receive SBRT to the gross tumor volume (GTV) at a dose of either 5Gy × 5-8 fractions or 4Gy × 15 fractions. After radiotherapy, participants will receive three cycles of tislelizumab (200mg Q3W) in combination with gemcitabine (1000mg/m² on Days 1 and 8) and cisplatin (25mg/m² on Days 1 and 8) or oxaliplatin (100mg/m² on Day 1), repeated every 21 days.

Patients will be re-evaluated after three cycles. If resectable, patients may undergo surgery, followed by additional postoperative therapy based on MDT recommendations. If unresectable, an additional three cycles of systemic therapy will be administered. The primary endpoint is overall survival (OS). Secondary endpoints include R0 resection rate, pathological complete response (pCR), surgical difficulty, local control rate, progression-free survival (PFS), and treatment-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, histologically or cytologically confirmed hilar cholangiocarcinoma
* Borderline resectable or unresectable disease based on imaging and MDT evaluation
* ECOG performance status 0-1
* Adequate hematologic, hepatic, and renal function
* No prior anti-tumor therapy for current diagnosis
* Expected survival ≥ 3 months
* Signed informed consent

Exclusion Criteria:

* Evidence of distant metastasis
* Prior treatment with immune checkpoint inhibitors
* Uncontrolled infection or serious medical comorbidities
* Active autoimmune disease requiring systemic therapy
* History of organ transplantation or immunodeficiency
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 36 months
  Defined as the time from initiation of treatment to death from any cause.

SECONDARY OUTCOMES:
R0 Resection Rate | At the time of surgery (approx. 3-6 months from enrollment)
  Proportion of patients achieving microscopically margin-negative (R0) resection among those undergoing surgery.
Pathological Complete Response (pCR) | At the time of surgery
  Absence of residual viable tumor cells in resected specimens.
Progression-Free Survival (PFS) | Up to 24 months
  Time from initiation of treatment to disease progression or death from any cause.
Local Control Rate | 6, 12, 18, and 24 months
  Proportion of patients without local tumor progression at irradiated site.
Treatment-related Adverse Events | From treatment initiation up to 90 days after last dose
  Frequency and severity of adverse events graded by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Principal Investigator — Shandong Cancer Hospital and Institute; Bo Zhang, Study Chair — Shandong Cancer Hospital and Institute